CLINICAL TRIAL: NCT04687306
Title: Inter-observer Reliability of Sacral Slope, Pelvic Femoral Motion and Cup Ante-inclination on Anteroposterior Pelvic Radiographs in Healthy Individuals.
Brief Title: Reliability of Sacral Slope, Pelvic Femoral Motion and Cup Ante-inclination on AP Pelvic Radiographs in Healthy Pts
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0719-20-FB
Record Dates: First submitted 2020-12-02; First posted 2020-12-29 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Females: 15 females
  Interventions: Diagnostic Test: X-rays- total of 4
- Males: 15 Males
  Interventions: Diagnostic Test: X-rays- total of 4

INTERVENTIONS:
Diagnostic Test: X-rays- total of 4 — X-rays of the sacral scope, pelvic femoral angle and cup ante-inclination in both sitting and standing positions

SUMMARY:
Currently, there are no validated anatomical landmarks that can be used to predict risk of and diagnose abnormal patterns of pelvic motion.This proposed study will measure sacral slope, pelvic femoral angle and cup ante-inclination in both sitting and standing positions, using healthy individuals without a history of spinal and/or lower extremity pathology. All radiographs will be evaluated for the three measurements by four individuals with the intent of evaluating inter-observer reliability. Determining the reproducibility of these angles between observers will give insight into the potential clinical utility of these measurements in evaluating and treating patients with hip-spine syndrome.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the mechanics and influence of spinopelvic motion and balance from normal healthy subjects for the purpose of establishing radiographic measurements which are reliable and reproducible and which could give insight into the potential clinical utility of these measurements as future predictors of who may/may not have spinal pelvic issues and in evaluation and treatment of patients with hip-spine syndrome.

This specific objective of this study will be to measure sacral slope, pelvic femoral angle and cup ante-inclination via radiographs in both sitting and standing positions. The radiographs will be evaluated for the three measurements by four individuals with the intent of evaluating inter-observer reliability.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals without major co-morbidities and without spine/hip/pelvis issues including previous injuries or surgeries

Exclusion Criteria:

* no history of spine/hip/pelvis issues
* females who are trying to get pregnant

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy individuals, both male and females aged 25-50 without major co-morbidities and without spine/hip/pelvis issues including previous injuries or surgeries
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Intraclass correlation coefficient (ICC) for Consistency in Spinopelvic Radiographic Measurements. | One year
  The intraclass correlation coefficient (ICC) will be used to evaluate the consistency of the 4 providers in measuring the sacral slope, pelvic femoral angle and cup ante-inclination via radiographs in both sitting and standing positions.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin L Garvin, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No